CLINICAL TRIAL: NCT06362551
Title: Retrospective Analysis of Differences in Information Provided by Donor Applicants Obtained by Written Application Compared to Genetic Risk Assessment Performed by Certified Genetic Counselor as Part of Routine Screening Process
Brief Title: Oocyte Donor Application Discrepancies
Status: Completed | Type: Observational
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Collaborators: GeneScreen Counseling, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: INC-GS-2024-002
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective observational study comparing information received on Inception Central Donor Recruitment's standardized online egg donor application compared to information reported during a Genetic Risk Assessment (GRA) consultation with a certified genetic counselor with contracted third party genetic counseling service, GeneScreen. All donor applicants completing a full application with Inception's Central Donor Recruitment and a GRA consultation with GeneScreen will be included.

DETAILED DESCRIPTION:
Background: Historically, it has been considered sufficient to have an egg donor applicant complete a written application that is reviewed by an egg donor program for acceptability. In 2021, ASRM put forth recommendations that "family history review and assessment of donors should be performed by a certified genetic counselor". In 2022, Inception Central Donor Recruitment (CDR) established a process for screening donor applicants that included Genetic Risk Assessment (GRA) with a certified genetic counselor. This study seeks to illustrate the discrepancies between personal and family history information documented on a standardized online application compared to a GRA consultation with a certified genetic counselor.

Objectives: Investigate the rate of new information obtained at GRA which was not included in the full application, as follows:

* New information with no change to health risk assessment (i.e. change in number of relatives)
* New information with a change to health risk assessment (i.e. known or suspected diagnoses for OD or family), with one of the following decisions

  * Still acceptable/approved for clinic (ie new multifactorial condition reported, such as diabetes)
  * Decline based on TPN internal guidelines alone (ie meets NCCN criteria for genetic testing)
  * Decline based on ASRM guidelines (ie first degree relative with a major malformation)

Hypothesis: Information obtained through GRA with a certified genetic counselor will lead to more detailed and accurate assessment of donor applicant eligibility. Some information obtained through GRA, which was not apparent on application, will lead to a donor applicant being declined based on internal Prelude Network Donor Screening Guidelines and/or guidelines set forth by the American Society of Reproductive Medicine.

ELIGIBILITY:
Inclusion Criteria:

* All oocyte donor applicants completing a full application with Inception's Central Donor Recruitment and a GRA consultation with GeneScreen will be included.

Exclusion Criteria:

* Not applicable

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Oocyte donors
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Rate of additional information | 6 months
  Simple statistical calculations will be evaluated for rate of additional information identified.
Rate of applicant decline | 6 months
  Simple statistical calculations will be evaluated for rate of applicant decline based on new information.

CONTACTS AND LOCATIONS:
Locations (1):
- Inception Fertility LLC, Houston, Texas, United States